CLINICAL TRIAL: NCT04206969
Title: Assessment of Transcultural Psychotherapy to Treat Major Depressive Disorder in Children and Adolescents From Migrant Families: a Bayesian Randomized Controlled Trial
Brief Title: Assessment of Transcultural Psychotherapy in Child Major Depressive Disorder
Acronym: EDPT-ADOS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: P180601; 2019-A01830-57 (Other: ID-RCB (ANSM))
Record Dates: First submitted 2019-12-16; First posted 2019-12-20 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Major Depressive Disorder
Keywords: Transcultural psychotherapy; migrant; child; adolescent; Depressive Disorder; psychiatric care; mixed studies; bayesian design; qualitative study; Randomized Controlled Trial
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcultural psychotherapy (Experimental): In addition to usual care, the participants in the treatment group receive transcultural psychotherapy in the inclusion centers, which consists of 5 sessions every 7 weeks (W6, W13, W20, W27, and W34). During all the research process, participants from both groups continue their usual care provided by the referent medical team outside the inclusion center.
  Interventions: Behavioral: Transcultural psychotherapy
- standard care (No Intervention): usual care provided by the referent medical team

INTERVENTIONS:
Behavioral: Transcultural psychotherapy — In addition to usual care, the participants receive transcultural psychotherapy
  Arms: Transcultural psychotherapy

SUMMARY:
The symptomatic and clinical expression of psychiatric disorders in children and adolescents is strongly influenced by the cultural setting they are growing up in. These cultural variations complicate psychiatric care, especially for migrant children, for whom appropriate care must be designed.

Transcultural psychotherapy is an original psychotherapeutic technique developed to meet these specific requirements in France and in different European and American countries. Its theoretical and methodological foundations rest on the works of George Devereux in ethnopsychiatry (1970). A psychotherapeutic technique intended for first-generation migrants was developed by Tobie Nathan and coll (1986). Marie-Rose Moro and colleagues (1990) have adapted this technique to second-generation migrants.

Indicated as a second-line treatment after the failure of standard management, this technique is fully formalized today. It comprises group consultations for the child and the family as a one-hour session each month, directed by a principal therapist, assisted by a group of co-therapists (of diverse cultural origins and occupations) and an interpreter in the family's mother tongue. The concept of culture is used to establish the therapeutic alliance, decode the symptoms, and propose treatment.

The children and adolescents receiving this treatment have varied psychopathological profiles, mostly involving depressive and/or anxiety disorders. Specifically, migrants' children are especially vulnerable to depression, their psychiatric care is generally longer and less effective than in the general population, and their rate of treatment failure higher.

Transcultural psychotherapy has demonstrated its value in these situations in numerous qualitative studies, but its efficacy has not yet been assessed by a method providing a high level of evidence, such as randomized controlled trials.

DETAILED DESCRIPTION:
Mixed method study using a multicenter, Bayesian randomized clinical trial with blinded evaluation of the primary outcome. Two parallel groups of 40 children or adolescents from 6 to 20 years-old and their family will be included. In the experimental group, patients will attend six sessions of transcultural therapy in addition to usual care. The improved Clinical Global Impression scale scores at 6 months will be compared across groups. Qualitative analysis of families and therapists' interviews will allow to specify the therapeutic processes and acceptability of the therapy.

ELIGIBILITY:
Inclusion Criteria:

* Be a child aged or an adolescent aged 6-20 years-old (this may be a declaratory age at the time of the consultation or based on a document for a residence request if no other identity documents are available)
* Be a first or second-generation migrant (born abroad or born from at least one parent who is born abroad)
* Have a psychological and/or psychiatric follow-up by a first-line care
* Have been referred for transcultural psychotherapy by their first line care to treat depression resistant to standard management.
* Present a depression according to the clinician who proposes the transcultural treatment (first line therapist), based on usual as well as cultural symptoms criteria of the below list:

  * Sadness
  * Diminish interest or pleasure in most of the usual activities
  * Insomnia or hypersomnia
  * Psychomotor agitation
  * Asthenia, loss of energy
  * Feeling of worthlessness or excessive guilt
  * Recurrent throughs of death
  * School problems (school failure, drop in grades, aggressivity with adult, school refusal…)
  * Mutism, and selective mutism
  * Runaways
  * Aggressivity
  * Impulsivity
  * Violence and delinquency
  * Conflicts with parents and adults from the community
  * Exclusion from family
  * Somatic pains
  * Massive separation anxiety
  * Regressive symptoms - loosing of an already acquired function such as speech, walk, stay alone for a sufficient time in relation to age, manage stress or anxiety for reasonable situations…
  * Denial of medical care for a chronic disease with no evident reasons
  * Cultural designation such as possessed by a spirit, being a child witch, or other cultural designations
  * State of trance The list is not exhaustive, and some other symptoms may be accepted if the first line clinician as well as the referent agree. The patients will be well characterized after inclusion.
* Present a score >= 4 on the iCGI - Severity at inclusion.
* Present transcultural issues confirmed by the referent (usual procedure of indirect pre-selection based on the presentation of the situation by referring physician)
* Have an informed consent signed by both parents/ one parent / tutor / adult patient (cf. 14.1 paragraph)

Exclusion Criteria:

* Patient or family has previously had transcultural psychotherapy
* Patient presents an acute psychiatric disorder which hinders the realization of the transcultural therapy - for example, excited delirium with great psychic disorganization, or high suicidal risk patients. These situations will be excluded during the screening time based on the first line therapist evaluation
* Patient presents an acute somatic disease which may hinder the well organization of the therapy
* Patient addressed for a legal expertise
* Child's/Adolescent's refusal
* Pregnant or breastfeeding (for women for young women of childbearing age)
* Participation in another interventional study
* Patient under guardianship or curatorship

Ages: 6 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-10-28 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Severity Score on the Improved Global Impression Scale (iCGI) to assess remission | at week 34 visit (v5)
  .iCGI score is a scale ranging from 1 to 7, 1 being Normal, not at all ill, and 7 - Among the most extremely ill patients.
  1. - Normal, not at all ill
  2. - Borderline mentally ill
  3. - Mildly ill
  4. - Moderately ill
  5. - Markedly ill
  6. - Severely ill
  7. - Among the most extremely ill patients
  Remission is defined as a mean iCGI score over the 3 experts <4 at 28 weeks of treatment (W34).

SECONDARY OUTCOMES:
Severity score on the iCGI | at baseline and weeks 6, 13, 20, 27 and 34 and 52
  To compare the course of the severity of depression in each group over the first 34 weeks after inclusion
Score on the French version of the Children's Depression Rating Scale-Revised (CDRS-R) | at baseline and weeks 6, 13, 20, 27 and 34 and 52
  It's a 17-item scale with answers on 5 or 7-point Likert scale (total score ranges from 17 to 113). A score ≥ 40 is indicative of depression, whereas a score ≤28 is often used to define remission.
  To compare the course of the level of depressive symptoms in each group over the first 34 weeks after inclusion
Score on the French version of the State-Trait Anxiety Inventory for children (STAI-C) | at baseline and weeks 6, 13, 20, 27 and 34 and 52
  To compare the course of the level of anxiety symptoms in each group over the first 34 weeks after inclusion
Score changes in Depression and anxiety Scores between Week 34 and week 52 | at 34 and 52 weeks
  To evaluate the persistence of the efficacy of transcultural psychiatry over time by describing the course of the severity of the depression and of the depressive and anxiety symptoms from 34 to 52 weeks after inclusion in the group of patients treated by transcultural psychotherapy during the first 34 weeks
analysis of the content of the clinical data collected during the visits | between 34 and 44 weeks
  To describe the therapeutic processes that enabled the improvement of patients treated by transcultural psychotherapy
analysis of the content of the interview with the families and therapists at the end of the treatment | between 34 and 44 weeks
  For this secondary objective concerning the group of patients treated by transcultural psychotherapy, a qualitative design will be used to explore the perceived efficacity and acceptability of the therapy. Investigators will organize two semi-structured interviews after the fifth therapy session. These semi-structured interviews will be conducted by a psychologist trained in transcultural care. One interview will concern the family and will explore, with the help of an interpreter speaking the native language of the family, the acceptability of the care as well as success factors identified by the family. The other interview will concern the therapists and will explore the success factors identified by the professionals. The interviews guides have been constructed by specialists of transcultural care in childhood and adolescence To describe the perceived efficacy and acceptability of the transcultural psychotherapy for the patient and the family

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan LACHAL, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (4):
- France (4):
  - Service de Psychopathologie de l'enfant, de l'adolescent, CHU Avicenne, Bobigny
  - Service de psychiatrie de l'enfant et de l'adolescent, CHRU Gabriel Montpied, Clermont-Ferrand
  - Maison de Solenn, Cochin Hospital, Paris
  - Centre Médico-psychologique, Service Universitaire de Psychiatrie de l'Enfant et de l'Adolescent, Hôpital La Grave, CHU Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No